CLINICAL TRIAL: NCT04063891
Title: Vibration Therapy as an Intervention for Enhancing Trochanteric Hip Fracture Healing in Elderly Patients: A Randomized Double-Blinded, Placebo-Controlled Clinical Trial
Brief Title: Vibration Therapy as an Intervention for Enhancing Trochanteric Hip Fracture Healing in Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince of Wales Hospital, Shatin, Hong Kong (Other)
Collaborators: Tai Po Hospital (Other Government)
Responsible Party: Principal Investigator, Ronald Man Yeung WONG, Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018.584
Record Dates: First submitted 2019-08-18; First posted 2019-08-21 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Hip Fractures
Keywords: Fracture healing, Osteoporosis, Vibration treatment
MeSH Terms: conditions — Hip Fractures; Osteoporosis

STUDY DESIGN:
Intervention Model Description: Randomized Double-Blinded, Placebo-Controlled Clinical Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo-Controlled (Placebo Comparator): Placebo group will have placebo treatment by standing on the LMHFV platform for 20 minutes/day
  Interventions: Device: Low-magnitude high-frequency vibration (LMHFV)
- Vibration Group (Experimental): Vibration group is treated with LMHFV at 35Hz, 0.3g, for 20 minutes/day, 5 times/week
  Interventions: Device: Low-magnitude high-frequency vibration (LMHFV)

INTERVENTIONS:
Device: Low-magnitude high-frequency vibration (LMHFV) — Low-magnitude high-frequency vibration (LMHFV) is a biophysical intervention that provides non-invasive, systemic mechanical stimulation and has been reported to have no adverse effect.
  Arms: Vibration Group
Device: Low-magnitude high-frequency vibration (LMHFV) — Placebo group will have sham treatment by standing on the LMHFV platform for 20 minutes/day
  Arms: Placebo-Controlled

SUMMARY:
Currently, there are approximately 300,000 hip fractures per year in the US with a mortality rate of 20% within 1 year. In Hong Kong, around 6,000 hip fractures occur yearly with costs approximately 52 million USD, and these numbers are projected to double by 2050.

The treatment of osteoporotic fractures is a major challenge as bone healing is delayed due to the impaired healing properties with respect to bone formation, angiogenesis and mineralization. Failure to unite results in pain, weakness, reduced mobility and fixation failure, and these complications are most common in elderly patients. Enhancement of osteoporotic fracture healing even after surgical fixation is therefore critical as a major goal in modern fracture management.

Low-magnitude high-frequency vibration (LMHFV) is a biophysical intervention that provides non-invasive, systemic mechanical stimulation and we are the first group to study its effect on fracture healing. Our previous animal studies have shown LMHFV to enhance healing from the early inflammation stage to the late phases of remodeling in osteoporotic diaphyseal fracture healing. Using our newly developed clinically relevant metaphyseal fracture model, we further proved the efficacy of LMHFV. Our results show LMHFV significantly enhanced fracture healing in both osteoporotic and normal rats radiologically by X-ray and micro-CT, histologically and biomechanically.

Justified with our preclinical studies, we hypothesize LMHFV can accelerate the time to fracture healing and enhance functional recovery. In this study, we propose to study the efficacy of LMHFV in trochanteric hip fracture healing by conducting a randomized double-blinded placebo-controlled clinical trial. Elderly patients aged 65 years or older of either gender, after surgical fixation, will be treated with LMHFV at 35Hz, 0.3g, 20 minutes/day, 5 days/week for 6 months. Results will be evaluated by clinical assessments, radiologically with X-rays, Computed Tomography (CT) and dynamic perfusion Magnetic Resonance Imaging (MRI) for blood circulation evaluation, Dual-energy X-ray absorptiometry (DXA), functional outcomes, and mortality. Positive findings from the study would have huge impact and change clinical practice.

DETAILED DESCRIPTION:
Osteoporosis predisposes patients to increased risk of fragility fractures, which affects clinical outcomes and functional recovery. In fact, the lifetime fracture risk of osteoporotic patients reaches as high as 40%. There are approximately 2.5 million osteoporotic fractures each year in the United States (US), with costs estimated at $15 billion USD in 2010. Currently, there are approximately 300,000 hip fractures per year in the US with a mortality rate of 20% within 1 year.

Low-magnitude high-frequency vibration (LMHFV) is a promising biophysical intervention that provides non-invasive, systemic mechanical stimulation. We previously conducted a randomized controlled trial with 710 healthy, active and independent postmenopausal women over 60 years old. The LMHFV group had significant improvements in reaction time, movement velocity, maximum excursion of balancing ability assessment and also quadriceps muscle strength (p<0.001). There were significantly lower fall incidences with 18.6% of 334 vibration group subjects compared with 28.7% of 327 control group subjects (adjusted HR=0.56, p=0.001). Benefits of LMHFV for balancing ability, muscle strength and risk of falling were retained 1 year after cessation of the treatment.

This is a randomized double-blinded placebo-controlled clinical trial to investigate the use of LMHFV to enhance trochanteric hip fracture healing and will provide impactful findings for the future management of osteoporotic fractures.

Objectives

1. To investigate the efficacy of LMHFV in trochanteric hip fractures on the time to radiological healing by conducting a randomized double-blinded placebo-controlled controlled clinical trial
2. To assess the effects of LMHFV in trochanteric hip fractures compared with control on clinical outcomes, densitometry, blood circulation, and mortality

Research Plan and Methodology A total of 120 unilateral trochanteric hip fracture (AO classification A1-A3) patients due to unintentional fall, aged 65 years or older, will be recruited. Patients will be randomized into either vibration or placebo group after surgical fixation with a cephalomedullary nail. Radiology will be taken after fixation and regular follow-up X-rays will be taken. CTs will also be taken to assess fracture healing. Blood circulation will be assessed by dynamic perfusion MR. BMD and Bone mineral content (BMC) at fracture site will be measured by Dual X-ray Absorptiometry (DXA) scan. Clinically, vital signs, wound condition and pain intensity will be monitored. Functional outcomes including Short Form-36 (SF-36), muscle strength, Timed up and go (TUG) test and balancing ability are evaluated. Mortality will be documented. Throughout the study, complications and safety issues will be documented and in case adverse events occur, treatment will be terminated immediately. The above parameters will be compared between pre- and post-treatment and between the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

1. Elderly male or females aged 65 years or older
2. Unilateral trochanteric hip fractures (AO classification A1-A3)
3. Due to unintentional fall
4. Fractures fixed with cephalomedullary nail (Gamma nail, Stryker - usual practise at our unit)
5. Willing and able to comply with study protocol

Exclusion Criteria:

1. Open fracture
2. Bilateral fractures
3. Patient with multiple injuries
4. Pathological fractures e.g. tumour, infection, etc.
5. History of medication or disease affecting bone metabolism such as hypo/hyperthyroidism, hypo/hyperparathyroidism, etc.
6. Malignancy
7. Chairbound or bedbound (unable to comply for LMHFV therapy)
8. Cognitive problems e.g. dementia (unable to agree for consent)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 83 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Change in time to healing | X-ray: baseline, 12, 52 weeks post-operation
  X-ray
Change in time to healing | 6 weeks post-operation
  Computed Tomography

SECONDARY OUTCOMES:
Densitometry | baseline, 6, 12 and 26 weeks post-operation
  Bone Mineral Density
Densitometry | baseline, 6, 12 and 26 weeks post-operation
  Bone mineral content
Blood circulation at fracture site | 6 weeks post-operation
  Measured by dynamic contrast-enhanced MR imaging
Pain scale | 2, 6, 12, 16, 20, 26, 36, 52 weeks post-operation
  Verbal Descriptor Scale (Pain Thermometer): scale ranges from 0 to 10, higher score indicates more pain
Quality of life questionnaire (SF-36) | 2, 6, 12, 16, 20, 26, 36, 52 weeks post-operation
  Functional status questionnaire to measure health-related quality of life in eight domains (physical functoning, physicial and emotional limitations, social functioning, bodily pain, general and mental health; Scores ranges from 0-100, higher score indicates better result.
Quadriceps muscle strength | 2, 6, 12, 16, 20, 26, 36, 52 weeks post-operation
  Dynamometer
Balancing ability | 2, 6, 12, 16, 20, 26, 36, 52 weeks post-operation
  Basic Balance Master System
Time up and go test (TUG) | 2, 6, 12, 16, 20, 26, 36, 52 weeks post-operation
  The subject will stand from a chair, walk 3 meters and travel back and sit back on the chair. The time is recorded
Mortality | 1 month, 3 months and 1 year post-operation

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Man Yeung Wong, MRCSEd, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Ronald Man Yeung Wong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rachner TD, Khosla S, Hofbauer LC. Osteoporosis: now and the future. Lancet. 2011 Apr 9;377(9773):1276-87. doi: 10.1016/S0140-6736(10)62349-5. Epub 2011 Mar 28. PMID 21450337
- [Background] Solomon DH, Patrick AR, Schousboe J, Losina E. The potential economic benefits of improved postfracture care: a cost-effectiveness analysis of a fracture liaison service in the US health-care system. J Bone Miner Res. 2014 Jul;29(7):1667-74. doi: 10.1002/jbmr.2180. PMID 24443384
- [Background] Black DM, Rosen CJ. Postmenopausal Osteoporosis. N Engl J Med. 2016 May 26;374(21):2096-7. doi: 10.1056/NEJMc1602599. No abstract available. PMID 27223157
- [Background] Shi HF, Cheung WH, Qin L, Leung AH, Leung KS. Low-magnitude high-frequency vibration treatment augments fracture healing in ovariectomy-induced osteoporotic bone. Bone. 2010 May;46(5):1299-305. doi: 10.1016/j.bone.2009.11.028. Epub 2009 Dec 2. PMID 19961960
- [Background] Bow CH, Tsang SW, Loong CH, Soong CS, Yeung SC, Kung AW. Bone mineral density enhances use of clinical risk factors in predicting ten-year risk of osteoporotic fractures in Chinese men: the Hong Kong Osteoporosis Study. Osteoporos Int. 2011 Nov;22(11):2799-807. doi: 10.1007/s00198-010-1490-0. Epub 2011 Jan 14. PMID 21234548
- [Background] Cheung WH, Sun MH, Zheng YP, Chu WC, Leung AH, Qin L, Wei FY, Leung KS. Stimulated angiogenesis for fracture healing augmented by low-magnitude, high-frequency vibration in a rat model-evaluation of pulsed-wave doppler, 3-D power Doppler ultrasonography and micro-CT microangiography. Ultrasound Med Biol. 2012 Dec;38(12):2120-9. doi: 10.1016/j.ultrasmedbio.2012.07.025. Epub 2012 Oct 11. PMID 23062367
- [Background] Leung KS, Yuen WF, Ngai WK, Lam CY, Lau TW, Lee KB, Siu KM, Tang N, Wong SH, Cheung WH. How well are we managing fragility hip fractures? A narrative report on the review with the attempt to setup a Fragility Fracture Registry in Hong Kong. Hong Kong Med J. 2017 Jun;23(3):264-71. doi: 10.12809/hkmj166124. Epub 2017 May 5. PMID 28473651
- [Background] Leung KS, Shi HF, Cheung WH, Qin L, Ng WK, Tam KF, Tang N. Low-magnitude high-frequency vibration accelerates callus formation, mineralization, and fracture healing in rats. J Orthop Res. 2009 Apr;27(4):458-65. doi: 10.1002/jor.20753. PMID 18924140
- [Background] Chung SL, Leung KS, Cheung WH. Low-magnitude high-frequency vibration enhances gene expression related to callus formation, mineralization and remodeling during osteoporotic fracture healing in rats. J Orthop Res. 2014 Dec;32(12):1572-9. doi: 10.1002/jor.22715. Epub 2014 Aug 17. PMID 25131218
- [Background] Chow DH, Leung KS, Qin L, Leung AH, Cheung WH. Low-magnitude high-frequency vibration (LMHFV) enhances bone remodeling in osteoporotic rat femoral fracture healing. J Orthop Res. 2011 May;29(5):746-52. doi: 10.1002/jor.21303. Epub 2010 Dec 23. PMID 21437955
- [Background] Wei FY, Chow SK, Leung KS, Qin J, Guo A, Yu OL, Li G, Cheung WH. Low-magnitude high-frequency vibration enhanced mesenchymal stem cell recruitment in osteoporotic fracture healing through the SDF-1/CXCR4 pathway. Eur Cell Mater. 2016 May 24;31:341-54. doi: 10.22203/ecm.v031a22. PMID 27215741
- [Background] Leung KS, Li CY, Tse YK, Choy TK, Leung PC, Hung VW, Chan SY, Leung AH, Cheung WH. Effects of 18-month low-magnitude high-frequency vibration on fall rate and fracture risks in 710 community elderly--a cluster-randomized controlled trial. Osteoporos Int. 2014 Jun;25(6):1785-95. doi: 10.1007/s00198-014-2693-6. Epub 2014 Mar 28. PMID 24676848
- [Background] Cheung WH, Li CY, Zhu TY, Leung KS. Improvement in muscle performance after one-year cessation of low-magnitude high-frequency vibration in community elderly. J Musculoskelet Neuronal Interact. 2016 Mar;16(1):4-11. PMID 26944817
- [Background] Griffith JF. Functional imaging of the musculoskeletal system. Quant Imaging Med Surg. 2015 Jun;5(3):323-31. doi: 10.3978/j.issn.2223-4292.2015.03.07. PMID 26029633
- [Background] Griffith JF, Genant HK. New imaging modalities in bone. Curr Rheumatol Rep. 2011 Jun;13(3):241-50. doi: 10.1007/s11926-011-0174-x. PMID 21369797
- [Background] Leung KS, So WS, Shen WY, Hui PW. Gamma nails and dynamic hip screws for peritrochanteric fractures. A randomised prospective study in elderly patients. J Bone Joint Surg Br. 1992 May;74(3):345-51. doi: 10.1302/0301-620X.74B3.1587874.
- [Background] Leung KS, Lee WS, Tsui HF, Liu PP, Cheung WH. Complex tibial fracture outcomes following treatment with low-intensity pulsed ultrasound. Ultrasound Med Biol. 2004 Mar;30(3):389-95. doi: 10.1016/j.ultrasmedbio.2003.11.008. PMID 15063521
- [Background] Herr KA, Garand L. Assessment and measurement of pain in older adults. Clin Geriatr Med. 2001 Aug;17(3):457-78, vi. doi: 10.1016/s0749-0690(05)70080-x. PMID 11459715
- [Background] Lisk R, Yeong K. Reducing mortality from hip fractures: a systematic quality improvement programme. BMJ Qual Improv Rep. 2014 Sep 19;3(1):u205006.w2103. doi: 10.1136/bmjquality.u205006.w2103. eCollection 2014. PMID 27493729
- [Background] Lau PY. To improve the quality of life in elderly people. Hong Kong Med J. 2016 Feb;22(1):4-5. doi: 10.12809/hkmj154782. No abstract available. PMID 26845466
- [Background] Chow SK, Chim YN, Wang J, Zhang N, Wong RM, Tang N, Leung KS, Cheung WH. Vibration treatment modulates macrophage polarisation and enhances early inflammatory response in oestrogen-deficient osteoporotic-fracture healing. Eur Cell Mater. 2019 Nov 7;38:228-245. doi: 10.22203/eCM.v038a16. PMID 31697398
- [Background] Wong RMY, Ho WT, Tang N, Tso CY, Ng WKR, Chow SK, Cheung WH. A study protocol for a randomized controlled trial evaluating vibration therapy as an intervention for postural training and fall prevention after distal radius fracture in elderly patients. Trials. 2020 Jan 16;21(1):95. doi: 10.1186/s13063-019-4013-0. PMID 31948477
- [Background] Rosso F, Dettoni F, Bonasia DE, Olivero F, Mattei L, Bruzzone M, Marmotti A, Rossi R. Prognostic factors for mortality after hip fracture: Operation within 48 hours is mandatory. Injury. 2016 Oct;47 Suppl 4:S91-S97. doi: 10.1016/j.injury.2016.07.055. Epub 2016 Aug 18. PMID 27546722
- [Background] Leung KS, Ko P. Practical manual for musculoskeletal trauma: Springer verlag; 2001.
- [Derived] Wong RMY, Wong PY, Liu C, Chui CS, Liu WH, Tang N, Griffith J, Zhang N, Cheung WH. Vibration therapy as an intervention for trochanteric hip fractures - A randomized double-blinded, placebo-controlled trial. J Orthop Translat. 2025 Jan 25;51:51-58. doi: 10.1016/j.jot.2025.01.002. eCollection 2025 Mar. PMID 39926341
- [Derived] Wong RMY, Chow SKH, Tang N, Chung YL, Griffith J, Liu WH, Ng RWK, Tso CY, Cheung WH. Vibration therapy as an intervention for enhancing trochanteric hip fracture healing in elderly patients: a randomized double-blinded, placebo-controlled clinical trial. Trials. 2021 Dec 4;22(1):878. doi: 10.1186/s13063-021-05844-y. PMID 34863272